CLINICAL TRIAL: NCT00190515
Title: Randomized Phase III Trial Comparing Adjuvant Oral UFT/LV to 5-FU/l-LV in Stage III Colorectal Cancer (JCOG-0205-MF)
Brief Title: A Trial Comparing Adjuvant Oral UFT/LV to 5-FU/l-LV in Stage III Colorectal Cancer (JCOG-0205-MF)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Haruhiko Fukuda (Other)
Collaborators: Ministry of Health, Labour and Welfare, Japan (Other Government)
Responsible Party: Sponsor-Investigator, Haruhiko Fukuda, JCOG Data Center, Japan Clinical Oncology Group
Organization: Japan Clinical Oncology Group (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JCOG-0205-MF; C000000193
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Colorectal Neoplasms
Keywords: adjuvant chemotherapy; Stage III colorectal cancer; 5-FU+l-LV; UFT+LV; randomized controlled trial
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): 5-FU/l-LV
  Interventions: Drug: 5FU+l-leucovorin
- 2 (Experimental): UFT/LV
  Interventions: Drug: UFT+Leucovorin

INTERVENTIONS:
Drug: 5FU+l-leucovorin — 5FU+l-leucovorin
  Arms: 1
Drug: UFT+Leucovorin — UFT+Leucovorin
  Arms: 2

SUMMARY:
To evaluate the clinical effectiveness of oral UFT/LV comparing 5-FU/l-LV as adjuvant therapy for stage III colorectal cancer.

DETAILED DESCRIPTION:
Oral fluoropyrimidines are widely used in practice for postoperative adjuvant chemotherapy for curatively resected colorectal cancer in Japan. In order to evaluate a clinical benefit of oral anticancer drugs in adjuvant chemotherapy, we conducted randomized controlled trial comparing the oral combination chemotherapy, UFT+LV, to the standard intravenous combination chemotherapy, 5-FU+l-LV, in stage III colorectal cancer.

UFT+LV: UFT 300mg/m2/day and LV 75mg/day, orally for 28days with 7days rest, repeated five times every 5 weeks.

5-FU+l-LV: 5-FU 500mg/m2, l-LV 250mg/m2, weekly administration for 6 times, repeated three times every 8 weeks.

Primary endpoints are disease-free survival and secondary endpoints are overall survival and adverse event rate.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically proved colorectal cancer (either adenocarcinoma, mucinous carcinoma, or signet-ring cell carcinoma).
2. Tumor is mainly located in between cecum and upper rectum, excluding that invades to lower rectum.
3. Stage III cancer by General Rules for Clinical and Pathological Studies on Cancer of the Colon, Rectum and Anus (6th ed.), excluding si(ai), n(-), M(-).
4. No synchronous colorectal cancer which invade muscularis propria or deeper.
5. Tumor resection with D2 or D3 lymph node dissection was performed.
6. Pathological determination of curability of tumor resection is cur A.
7. Age at registration is above 20 and below 75 years old.
8. ECOG Performance status is 0 or 1.
9. No prior chemotherapy or radiation therapy.
10. Intake of normal diet and oral drugs is possible.
11. Major organ function is preserved. WBC>=3,000/mcl, PLT>=100,000/mcl, GOT<=100 IU/L, GPT<=100 IU/L, T.Bil <=2.0 mg/dl, Cr<=1.5 mg/dl
12. Adjuvant chemotherapy can be started within 9 weeks after surgery.
13. Written informed consent is taken.

Exclusion Criteria:

1. Active co-existing malignancy （synchronous or metachronous malignancy whose disease free period is within 5 years). Carcinoma in situ is eligible.
2. Severe postoperative complications which do not resolve until registration.
3. There is following complication. insulin-controlling or uncontrollable diabetes mellitus, uncontrollable hypertension, myocardial infarction within six month or unstable angina pectoris, liver cirrhosis, interstitial pneumonia, pulmonary fibrosis, severe emphysema
4. Pregnant or breast-feeding woman.
5. Difficult to participate with the trial, having mental disorder or psychiatric symptoms.
6. Judged to be inappropriate to register.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1101 (Actual)
Dates: Start 2003-02; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Disease-free survival | during the study conduct

SECONDARY OUTCOMES:
Overall survival | during the study conduct
Rate of adverse event | during the study conduct

CONTACTS AND LOCATIONS:
Overall Officials: Yoshihiro Moriya, MD, Study Chair — National Cancer Center Hospital
Locations (48):
- Japan (48):
  - Aichi Cancer Center Hospital, Nagoya,Chikusa-ku,Kanokoden,1-1, Aichi-ken
  - Fujita Health University, Toyoake,Kutsukake-cho,Dengakugakubo,1-98, Aichi-ken
  - Chiba Cancer Center Hospital, Chiba,Chuo-ku,Nitona-cho,666-2, Chiba
  - National Cancer Center Hospital East, Kashiwa,Kashiwanoha,6-5-1, Chiba
  - Toho University Sakura Hospital, Sakura,Shimoshidu,564-1, Chiba
  - Jyuntendo Urayasu Hospital, Urayasu,Tomioka,2-1-1, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama,Horinouchi,13, Ehime
  - National Kyushu Cancer Center, Fukuoka,Minami-ku,Notame,3-1-1, Fukuoka
  - Kurume University School of Medicine, Kurume,Asahi-machi,67, Fukuoka
  - Kurume University Medical Center, Kurume,Kokubumachi,155-1, Fukuoka
  - Gunma Prefectural Cancer Center, Ota,Takabayashi-nishi-cho,617-1, Gunma
  - Hiroshima University, School of Medicine, Hiroshima,Minami-ku,Kasumi,1-2-3, Hiroshima
  - Hiroshima City Hospital, Hiroshima,Naka-ku,Motomachi,7-33, Hiroshima
  - Sapporo-Kosei General Hospital, North-3,East8-5,Chuou-ku,Sapporo, Hokkaido
  - Kansai Rosai Hospital, Amagasaki,Inabasou,3-1-69, Hyōgo
  - Ibaraki Kenritsu Chuo Hospital & Cancer Center, Nishi-ibarakigun,Tomobemachi,Koibuchi,6528, Ibaraki
  - Ishikawa Prefectual Central Hospital, Kanazawa,Kuratsuki-Higashi,2-1, Ishikawa-ken
  - Teikyo University Hospital, Mizonokuchi, Kawasaki,Takatsu-ku,Mizonokuchi,3-8-3, Kanagawa
  - Kitasato University East Hospital, Sagamihara,Asamizodai,2-1-1, Kanagawa
  - Kitasato University School of Medichine, Sagamihara,Kitasato,1-15-1, Kanagawa
  - Yokohama City University Medical Center, Yokohama,Minami-ku,Urafunecho,4-57, Kanagawa
  - Kanagawa Cancer Center, Yokohama,Nakao,Asahi-ku,1-1-2, Kanagawa
  - Showa University Northern Yokohama Hospital, Yokohama,Tsuzuki-ku,Chigasakichuo,35-1, Kanagawa
  - National Hospital Organization Kyoto Medical Center, Kyoto,Fushimi-ku,Fukakusa,Mukaihata-cho,1-1, Kyoto
  - Miyagi Cancer Center, Natori,Medeshima-Shiode,Nodayama,47-1, Miyagi
  - Nagano Municipal Hospital, Nagano,Tomitake,1333-1, Nagano
  - Niigata Cancer Center Hospital, Niigata,Kawagishi-cho,2-15-3, Niigata
  - Oita University Fuculty of Medicine, Oita,Hasama-machi,Oogaoka,1-1, Oita Prefecture
  - Okayama Saiseikai General Hospital, Okayama,Ifukucho,1-17-18, Okayama-ken
  - Minoh City Hospital, Minoh,Kayano,5-7-1, Osaka
  - Osaka National Hospital, Osaka,Chuo-ku,Hoenzaka,2-1-14, Osaka
  - Osaka Medical Center for Cancer and Cardiovascular Diseases, Osaka,Higashinari-ku,Nakamichi,1-3-3, Osaka
  - Osaka City General Hospital, Osaka,Miyakojima-ku,Miyakojimahondori,2-13-22, Osaka
  - Sakai Municipal Hospital, Sakai,Minamiyasuicho,1-1-1, Osaka
  - Osaka University Graduate School of Medicine, Suita,Yamada-oka,2-2, Osaka
  - Osaka Medical College, Takatsuki,Daigakucho,2-7, Osaka
  - Omiya Medical Center, Jichi Medical School, Saitama,Omiya-ku,Amanuma-cho,1-847, Saitama
  - National Defense Medical College, Tokorozawa,Namiki,3-2, Saitama
  - Sizuoka Cancer Center, Sunto-gun,Nagaizumi-cho,Shimonagakubo,1007, Shizuoka
  - Tochigi Cancer Center, Utsunomiya,Yohnan,4-9-13, Tochigi
  - Tokyo Medical and Dental University Hospital, Bunkyo-ku,Yushima,1-5-45, Tokyo
  - National Cancer Center Hospital, Chuo-ku, Tsukiji, 5-1-1, Tokyo
  - Toho University Ohashi Hospital, Meguro-ku,Ohashi,2-17-6, Tokyo
  - Toranomon Hospital, Minato-ku,Toranomon,2-2-2, Tokyo
  - Kyorin University School of Medicine, Mitaka,Shinkawa,6-20-2, Tokyo
  - Tokyo Medical University, Shinjuku-ku,Nishi-shinjuku,6-7-1, Tokyo
  - Keio University Hospital, Shinjuku-ku,Shinanomachi,35, Tokyo
  - Yamagata Prefectural Central Hospital, Yamagata,Aoyagi,1800, Yamagata

REFERENCES:
- See also: Related Info — http://www.jcog.jp/